CLINICAL TRIAL: NCT07326215
Title: A Study of the Efficacy and Safety of Extracorporeal Carbon Dioxide Removal Using PrismaLung+ in Chinese Critically Ill Patients: a Prospective Randomized Controlled Clinical Trial
Brief Title: A Study of the Efficacy and Safety of Extracorporeal Carbon Dioxide Removal Using PrismaLung+
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Vantive Health LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BXU614243
Record Dates: First submitted 2025-12-09; First posted 2026-01-08 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2025-12

CONDITIONS: Acute Respiratory Distress Syndrome; Acute Kidney Injury
MeSH Terms: conditions — Respiratory Distress Syndrome; Acute Kidney Injury

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients receiving IMV combined with ECCO2R (Experimental): Patients will receive IMV combined with ECCO2R using PrismaLung+.
  Interventions: Device: PrismaLung+
- Patients receiving IMV alone (Active Comparator)
  Interventions: Other: Invasive Mechanical Ventilation

INTERVENTIONS:
Device: PrismaLung+ — PrismaLung+ is a medical device that provides ECCO2R as a stand-alone therapy or in combination with CRRT. The planned treatment duration with PrismaLung+ for patients in the study group is 7 days. However, the Investigator can discontinue PrismaLung+ treatment before 7 days if ECCO2R is no longer required. Following the 7-day treatment period, the Investigator will assess the patient's condition to determine whether to continue ECCO2R. Patients will require systemic anticoagulation with heparin during ECCO2R treatment.
  Continuous renal replacement therapy may be administered concurrently to patients during the study, if needed, at the discretion of the Investigator. During the study, patients will be given active treatment for their primary disease.
  Arms: Patients receiving IMV combined with ECCO2R
Other: Invasive Mechanical Ventilation — According to the standard clinical practice of IMV, oral or nasal endotracheal intubation can be used for IMV. The initial mode of IMV and ventilatory parameters will be determined based on the patient's condition, and an appropriate patient-centered LPV approach will be selected to adjust the ventilatory parameters to achieve the study LPV strategy. Appropriate treatments other than ECCO2R will be provided for this group. Continuous renal replacement therapy may be administered concurrently to patients during the study, if needed, at the discretion of the Investigator. During the study, patients will be given active treatment for their primary disease.
  Arms: Patients receiving IMV alone

SUMMARY:
PrismaLung+ is a sterile, single-use medical device aimed at performing partial removal of carbon dioxide (CO2) from the patient's venous blood via diffusion through a membrane. The goal of this prospective, open label, randomized controlled study is to evaluate the efficacy and safety of PrismaLung+ on extracorporeal carbon dioxide removal (ECCO2R) in critically ill patients under invasive mechanical ventilation (IMV). Patients will be randomized to receive either IMV combined with ECCO2R (using PrismaLung+) in the study group or IMV alone in the control group, at a ratio of 2:1.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years old.
2. Invasive mechanical ventilation patients with PaCO2 > 50 mmHg and pH < 7.4 under LPV strategy (RR < 25/min, DP < 15 cmH2O).
3. Expected to be able to tolerate ECCO2R for a minimum of 2h.
4. Patients signed a written informed consent; if the right to consent cannot be exercised due to loss of decision-making ability or impairment of consciousness, the legal representative or immediate family member must sign the informed consent document after fully understanding the research content.

Exclusion Criteria:

1. Body weight < 30 kg.
2. Has a contraindication for systemic anticoagulation with heparin according to the Investigator.
3. Patient unable to establish extracorporeal circulation access or has a high risk of establishing such access, as judged by the Investigator.
4. Allergic to the investigational device/tubing, and/or to the CRRT filters/tubing if combined with CRRT treatment.
5. Expected to require extracorporeal membrane oxygenator (ECMO) treatment within 24h after enrollment.
6. Patient's primary disease is expected to worsen rapidly or require other surgical intervention within 24h after enrollment.
7. Diagnosed as brain dead or in a vegetative state.
8. Pregnant and/or breastfeeding.
9. Plans to participate in other device studies within 30 days before screening or during the study period or has completed any clinical drug study within 5 half lives of the investigational drug.
10. Patients is considered as unsuitable for participating in the study, as judged by the Investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 99 (Estimated)
Dates: Start 2025-12-31 (Estimated); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
The percent decrease of partial pressure of carbon dioxide (PaCO2) from baseline after 2h of treatment. | 2 hours after treatment
  Percent decrease (%) of PaCO2 from baseline based on arterial blood gas 2h after treatment initiation.
  Must meet the following requirements for data collection:
  1. maintained LPV (RR < 25/min, DP < 15 cmH2O) with consistent ventilatory parameters with baseline;
  2. blood flow rate (Qb) of 300 to 450 mL/min;
  3. sweep gas flow rate of 10 L/min.

SECONDARY OUTCOMES:
CO2 clearance (in the experimental group only) | 2 hours and 24 hours after treatment
  Blood sampled pre- and post-PrismaLung+ filter to calculate CO2 clearance based on blood gas analysis results.
Changes in Blood Gas Indexes | 2 hours, 4 hours, 8 hours, 12 hours, 24 hours, 2 days, 3 days, 7 days after treatment
  Change in blood gas indexes before and after treatment based on arterial blood gas at different follow-up timepoints. Blood gas indexes include pH, PaO2, PaCO2, SaO2, standard bicarbonate (SB), actual bicarbonate (AB), and lactic acid.
Changes in Oxygenation Indexes (PaO2/FiO2) | 2 hours, 4 hours, 8 hours, 12 hours, 24 hours, 2 days, 3 days, 7 days after treatment
  The ratio of partial pressure of arterial oxygen (PaO2 in mmHg) to fraction of inspired oxygen (FiO2 in %), i.e., PaO₂/FiO₂.
Changes in Ventilatory Parameters | 2 hours, 4 hours, 8 hours, 12 hours, 24 hours, 2 days, 3 days, 7 days after treatment
  Changes in respiratory rate (RR). The following definitions on ventilatory parameters are for reference and the specific parameters are based on the ventilator mode at each site.
  RR refers to the number of breaths per minute of a ventilator, measured in breaths/min.
Changes in Ventilatory Parameters | 2 hours, 4 hours, 8 hours, 12 hours, 24 hours, 2 days, 3 days, 7 days after treatment
  Changes in tidal volume (VT). The following definitions on ventilatory parameters are for reference and the specific parameters are based on the ventilator mode at each site.
  VT refers to the volume of air delivered by a ventilator, measured in mL.
Changes in Ventilatory Parameters | 2 hours, 4 hours, 8 hours, 12 hours, 24 hours, 2 days, 3 days, 7 days after treatment
  Changes in driving pressure (DP). The following definitions on ventilatory parameters are for reference and the specific parameters are based on the ventilator mode at each site.
  DP refers to the driving pressure of a respiratory system, defined as tidal volume/respiratory system compliance. Respiratory system driving pressure = airway Pplat - PEEP, measured in cmH2O.
Changes in Ventilatory Parameters | 2 hours, 4 hours, 8 hours, 12 hours, 24 hours, 2 days, 3 days, 7 days after treatment
  Changes in positive end-expiratory pressure (PEEP). The following definitions on ventilatory parameters are for reference and the specific parameters are based on the ventilator mode at each site.
  PEEP refers to the pressure applied by a ventilator that will remain in the airways at the end of exhalation, measured in cmH2O.
Changes in Ventilatory Parameters | 2 hours, 4 hours, 8 hours, 12 hours, 24 hours, 2 days, 3 days, 7 days after treatment
  Changes in plateau pressure (Pplat). The following definitions on ventilatory parameters are for reference and the specific parameters are based on the ventilator mode at each site.
  Pplat refers to the airway plateau pressure, i.e., the airway pressure when airflow has ceased or is paused at the end of inspiration, measured in cmH2O.
Changes in Ventilatory Parameters | 2 hours, 4 hours, 8 hours, 12 hours, 24 hours, 2 days, 3 days, 7 days after treatment
  Changes in fraction of inspired oxygen (FiO2). The following definitions on ventilatory parameters are for reference and the specific parameters are based on the ventilator mode at each site.
  FiO2 refers to the fraction of oxygen in the delivered gas under monitoring, measured in percentage.
Ventilator-Free Days | 28 days after enrollment
  The number of days between successful weaning from mechanical ventilation and the end of follow-up (28 days after treatment).
  Weaning from mechanical ventilation refers to the removal of mechanical ventilation for respiratory support and the resumption of complete spontaneous breathing, after the primary disease is controlled and the ventilation and gas exchange functions are improved in patients under mechanical ventilation (referred to as weaning from mechanical ventilation). Instead of using mechanical ventilation for respiratory support, the respiratory load of the body is borne entirely by the patient's own respiratory capacity.
  Spontaneous breathing:
  * The total respiratory rate of the patient is higher than that set in the assist-control mode during mechanical ventilation, or the mechanical ventilation mode requires the patient to breathe spontaneously.
  * No invasive respiratory support is provided.
Days of ICU stay | 28 days after enrollment
  The span of time during which the patient receives treatment and care in the ICU within 28 days after treatment initiation.
28-day mortality | 28 days after enrollment
  All-cause mortality and in-hospital mortality after enrollment.
Quality of life (QoL) | 1 day of regaining consciousness, 28 days after enrollment.
  During the trial, for patients who regain consciousness, the differences in quality-of-life scores will be evaluated based on EQ-5D-5L assessments at the time of awakening and on Day 28 (if the patients are still alive).

CONTACTS AND LOCATIONS:
Locations (10):
- China (10):
  - China-Japan Friendship Hospital, Beijing, Beijing Municipality
  - The First Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong
  - The University of Hong Kong-Shenzhen Hospital, Shenzhen, Guangdong
  - The First Affiliated Hospital of Harbin Medical University, Harbin, Heilongjiang
  - Zhongda Hospital Southeast University, Nanjing, Jiangsu
  - The First Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - ZhongShan Hospital Fudan University, Shanghai, Shanghai Municipality
  - Sichuan Provincial People's Hospital, Chengdu, Sichuan
  - The First Affiliated Hospital Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - Sir Run Run Shaw Hospital Zhejiang University School of Medicine, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No